CLINICAL TRIAL: NCT04837196
Title: A Phase 1/2, Open-label Study Investigating the Safety, Tolerability and Efficacy of ASP7517 as a Single Agent and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors Known to Express WT1 Antigen
Brief Title: Study of ASP7517 Alone and With Pembrolizumab in Participants With Advanced Solid Tumors Expressing WT1 Antigen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7517-CL-1101
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignancies; Advanced Cancer
Keywords: Solid Tumors; ASP7517; WT1 Antigen
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 cells/dose) (Experimental): Participants received one dose of ASP7517 1x10^7 cells/dose for up to 6 doses (168 days) by intravenous (IV) infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days). Following first 2 cycles, participants not meeting treatment discontinuation criteria and receiving clinical benefit (defined:radiological response/SD/reduction of disease-related symptoms) continued treatment with ASP7517. After 4 cycles of treatment, participants achieving confirmed CR discontinued ASP7517, and participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD and those not clinically stable or clinical progression was confirmed by investigator and followed up to 48 weeks until iCPD per independent central review, initiation of new anticancer therapy or meeting 1 of Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days.
  Interventions: Drug: ASP7517
- Phase 1: Monotherapy dose escalation (ASP7517 1x10^8 cells/dose) (Experimental): Participants received one dose of ASP7517 1x10^8 cells/dose by IV infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days). Following first 2 cycles, participants not meeting treatment discontinuation criteria and receiving clinical benefit (defined as radiological response/ SD, or reduction of disease-related symptoms) continued treatment with ASP7517. After 4 cycles of treatment, participants achieving confirmed CR discontinued ASP7517, and any participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD and those not clinically stable or clinical progression was confirmed by the investigator and followed for up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days
  Interventions: Drug: ASP7517
- Phase 2:Monotherapy dose expansion (ASP7517 1x10^8 cells/dose) (Experimental): Participants received ASP7517 1x10^8 cells/dose by IV infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days).Following the first 2 cycles, participants not meeting discontinuation criteria and were receiving clinical benefit (defined as radiological response/SD, or reduction of disease-related symptoms) continued treatment with ASP7517. After 4 cycles of treatment, participants achieving confirmed CR discontinued ASP7517, and any participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD and who were not clinically stable or clinical progression was confirmed by the investigator and followed up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the EOT visit, participants completed the Safety follow-up visits 30, 60 and 90 days.
  Interventions: Drug: ASP7517
- Phase1:Combination Therapy dose Escalation (ASP7517 1x10^7 cells/dose) and Pembrolizumab (Experimental): Participants received ASP7517 1x10^7 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4-6 mL/min) (1 Cycle = 28 days) with 400 mg pembrolizumab infusion (over 30 min) for up to 4 doses every 6 weeks. After 2 cycles, those not meeting discontinuation criteria and receiving clinical benefit continued ASP7517 and pembrolizumab. Participants with confirmed CR within 4 cycles did not receive ASP7517 at cycles 5-6; those with PR/SD after 4 doses received 2 more ASP7517 doses with pembrolizumab. After Treatment Period, all except those with iCPD, iUPD, or clinical progression entered Observation Period and continued pembrolizumab alone (up to 17 doses) to monitor response up to 96 weeks until iCPD, new therapy, or discontinuation criteria. After EOT visit, participants completed Safety follow-up at 30, 60, and 90 days.
  Interventions: Drug: ASP7517; Drug: Pembrolizumab
- Phase 1:Combination Therapy dose Escalation (ASP7517 1x10^8cells/dose) and Pembrolizumab (Experimental): Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4-6 mL/min) (1 Cycle = 28 days) with 400 mg pembrolizumab infusion (over 30 min) for up to 4 doses every 6 weeks. After 2 cycles, those not meeting discontinuation criteria and receiving clinical benefit continued ASP7517 and pembrolizumab. Participants with confirmed CR within 4 cycles did not receive ASP7517 at cycles 5-6; those with PR/SD after 4 doses received 2 more ASP7517 doses with pembrolizumab. After Treatment Period, all except those with iCPD, iUPD, or clinical progression entered Observation Period and continued pembrolizumab alone (up to 17 doses) to monitor response up to 96 weeks until iCPD, new therapy, or discontinuation criteria. After EOT visit, participants completed Safety follow-up at 30, 60, and 90 days.
  Interventions: Drug: ASP7517; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ASP7517 — Intravenous (IV)
Drug: Pembrolizumab — Intravenous (IV)
  Arms: Phase 1:Combination Therapy dose Escalation (ASP7517 1x10^8cells/dose) and Pembrolizumab; Phase1:Combination Therapy dose Escalation (ASP7517 1x10^7 cells/dose) and Pembrolizumab

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and clinical response of ASP7517, and determine the Recommended Phase 2 Dose (RP2D) and/or the Maximum Tolerated Dose (MTD) of ASP7517 when administered as a single agent and in combination with pembrolizumab.

This study also evaluated other measures of anticancer activity of ASP7517 when administered as a single agent and in combination with pembrolizumab based on central and local assessment.

DETAILED DESCRIPTION:
This study consisted of arms receiving ASP7517 monotherapy and arms receiving ASP7517 and pembrolizumab combination therapy in Phase 1 (dose escalation cohort) and Phase 2 (dose expansion cohort). Phase 2 monotherapy and combination dose expansion cohorts were opened after the phase 1 escalation cohort was completed.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally-advanced (unresectable) or metastatic solid tumor malignancy that is confirmed by available pathology records or current biopsy. Participant must also have received all standard therapies (unless the therapy is contraindicated or intolerable) appropriate to provide clinical benefit for his/her specific tumor type. However, participants with metastatic melanoma who have not received checkpoint inhibitors [CPIs] (i.e., CPIs naive) may enroll in the Phase 2 Combination Therapy Arm Dose Expansion Cohort to receive CPI: Pembrolizumab.
* Participant must be diagnosed with solid tumor known to express WT1 antigen such as, but not limited to melanoma, ovarian cancer or Colorectal Cancer (CRC).
* Participant consents to provide an archival tumor specimen in a tissue block or unstained serial slides, if available, prior to study treatment.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Participant's last dose of prior antineoplastic therapy, including any immunotherapy, was 21 days or 5 half-lives, whichever is shorter, prior to initiation of IP administration. A participant with BRAF gene, epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation positive non-small cell lung carcinoma is allowed to remain on epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) or anaplastic lymphoma kinase (ALK) or BRAF inhibitor therapy until 4 days prior to the start of Investigational Product (IP) administration.
* Participant has completed any radiotherapy (including stereotactic radiosurgery) at least 2 weeks prior to IP administration.
* Participant's Adverse Events (AEs) (excluding alopecia) from prior therapy have improved to grade 1 or baseline within 14 days prior to start of IP.
* Participant has adequate organ function prior to start of IP. If a participant has received a recent blood transfusion, the laboratory tests must be obtained ≥ 4 weeks after any blood transfusion.
* A female participant is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after the final IP administration.
* Female participant must agree not to breastfeed starting at screening and throughout the IP and for 180 days after the final IP administration.
* Female participant must not donate ova starting at screening and throughout the IP and for 180 days after the final IP administration.
* A male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for at least 180 days after the final IP administration.
* Male participant must not donate sperm during the treatment period and for 180 days after the final IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 180 days after the final IP administration.
* Participant agrees not to participate in another interventional study while receiving IP.

Additional Inclusion Criteria for Participants in the Expansion Cohorts:

* Participant meets one of the following:

  * Participant has the tumor type for which a confirmed response was observed in a monotherapy dose escalation cohort (monotherapy arm only) cohort; OR
  * For tumor specific expansion cohorts of ASP7517 or ASP7517 with pembrolizumab, participant has the applicable tumor type; CPI refractory metastatic melanoma (monotherapy and combination arms), CPI naïve melanoma (combination arm only), ovarian cancer, colorectal cancer (CRC).
* Participant has at least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant consents to provide a tumor specimen in a tissue block or unstained serial slides obtained within 56 days prior to first dose of IP. If a recent tissue sample cannot be provided due to medical or safety concerns, enrollment into the study must be discussed with the medical monitor.
* Participant consents to undergoing a tumor biopsy (core tissue biopsy or excision) during the treatment period as indicated in the schedule of assessments if predose biopsy is available and if medically feasible.

Exclusion Criteria:

* Participant weighs < 45 kg at screening.
* Participant has received investigational therapy (other than an investigational EGFR TKI in a participant with EGFR activating mutations or ALK or BRAF inhibitor in a participant with an ALK mutation) within 21 days or 5 half-lives, whichever is shorter, prior to start of IP.
* Participant requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to Cycle 1 Day 1. Participants using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone up to 10 mg per day of prednisone) are allowed.
* Participant has symptomatic central nervous system (CNS) metastases or participant has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Participants with previously treated CNS metastases are eligible, if they are clinically stable and have no evidence of CNS progression by imaging for at least 4 weeks prior to start of IP and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone or > 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Participant has an active autoimmune disease. Participants with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy or skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
* Participant was discontinued from prior immunomodulatory therapy due to a grade ≥ 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Participant has known history of serious hypersensitivity reaction to a known ingredient of ASP7517 or pembrolizumab or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Participant has a known history of human immunodeficiency virus.
* Participant with known history of positive hepatitis B surface antigen or isolated hepatitis B core antibody (including acute HBV or chronic HBV) or hepatitis C ([HCV] ribonucleic acid [RNA] detected by qualitative assay). Hepatitis C RNA testing is not required in participants with negative hepatitis C antibody testing.
* Participant has received a live vaccine against infectious diseases within 28 days prior to initiation of IP.
* Participant has a history of drug-induced pneumonitis (interstitial lung disease), a history of (non-infectious) pneumonitis that required steroids, radiation pneumonitis or currently has pneumonitis.
* Participant has an infection requiring systemic therapy within 14 days prior to IP.
* Participant has received a prior allogeneic bone marrow or solid organ transplant.
* Participant is expected to require another form of antineoplastic therapy while on IP.
* Participant has had a myocardial infarction or unstable angina within 6 months prior to the start of IP or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant has a clinically significant abnormal electrocardiogram at screening.
* Participant has symptomatic cardiovascular disease within the preceding 12 months unless cardiology consultation and clearance has been obtained for study participation, including but not limited to the following: significant coronary artery disease (e.g., requiring angioplasty or stenting), acute myocardial infarction or unstable angina pectoris < 3 months prior screening, uncontrolled hypertension, clinically significant arrhythmia or congestive heart failure (New York Heart Association grade ≥ 3).
* Any condition that makes the participant unsuitable for study participation.
* Participant has had a major surgical procedure and has not completely recovered within 28 days prior to the start of IP.
* Participant has a prior malignancy active (i.e., requiring treatment of intervention) within the previous 2 years prior to the screening visit, except for locally curable malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast. Participants with organ confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been surgically removed or treated with definitive radiotherapy.
* Participant has International Normalized Ratio (INR) > 1.5 x Upper Limits of Normal (ULN) and/or activated partial thromboplastin time (aPTT) > 1.5 x institutional normal limits.

Additional Exclusion Criteria for Participants in Combination Expansion Cohorts:

* Participants with metastatic CRC with documented microsatellite instability-high (MSI-H) or mismatch repair (MMR) deficient who have received prior treatment with PD-1 or programmed death-ligand (PD-L1) inhibitors such as nivolumab or pembrolizumab.
* CPI naïve metastatic melanoma participants who have received PD-1 or PD-L1 inhibitors, such as nivolumab or pembrolizumab.
* Participants with metastatic ovarian cancer with documented MSI-H or MMR deficient who have received PD-1or PD-L1 inhibitors, such as nivolumab or pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals, Iowa City, Iowa
  - UPCI Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/7517-CL-1101
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14590&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged ≥ 18 years diagnosed with a locally-advanced (unresectable) or metastatic solid tumor known to express Wilms' tumor protein 1 (WT1) antigen were enrolled in this study.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study. No combination therapy dose expansion arm was enrolled.
Groups:
- Phase 1:Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose): Participants received one dose of ASP7517 1x10^7 cells/dose for up to 6 doses (168 days) by intravenous (IV) infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days). Following the first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (defined as radiological response or stable disease [SD], or reduction of disease-related symptoms) continued further treatment with ASP7517, as decided by the investigator. After completing 4 cycles of treatment, any participant who achieved confirmed complete response (CR) did not continue with ASP7517, and any participants who achieved partial response (PR) or SD received an additional 2 doses. Participants entered an Observation Period except those with "immune" confirmed progressive disease (iCPD), unconfirmed disease progression disease (iUPD) (per independent central review or local review) and who were not clinically stable or clinical progression was confirmed by the investigator and were followed for up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the end of treatment (EOT) visit, participants completed the Safety follow-up visits 30, 60 and 90 days.
- Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose): Participants received one dose of ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) by IV infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days). Following the first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (defined as radiological response or SD, or reduction of disease-related symptoms) continued further treatment with ASP7517, as decided by the investigator. After completing 4 cycles of treatment, any participants who achieved confirmed CR did not continue with ASP7517, and any participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD (per independent central review or local review) and who were not clinically stable or clinical progression was confirmed by the investigator and were followed for up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the EOT visit, participants completed the Safety follow-up visits 30, 60 and 90 days.
- Phase 2:Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose): Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) by IV infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days).Following the first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (defined as radiological response or SD, or reduction of disease-related symptoms) continued further treatment with ASP7517, as decided by the investigator. After completing 4 cycles of treatment, any participants who achieved confirmed CR did not continue with ASP7517, and any participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD (per independent central review or local review) and who were not clinically stable or clinical progression was confirmed by the investigator and were followed for up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the EOT visit, participants completed the Safety follow-up visits 30, 60 and 90 days.
- Phase 1:Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab: Participants received ASP7517 1x10^7 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4 to 6 mL/minute) (1 Cycle=28 days) in combination with 400mg pembrolizumab infusion (over 30 minutes) with up to 4 doses every 6 weeks. Following first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (defined as radiological response or SD, or reduction of disease-related symptoms) continued further treatment with ASP7517 and pembrolizumab as decided by the investigator. Participants who achieved confirmed CR within first 4 cycles could not receive further treatment with ASP7517 at cycle 5 and 6; and participants who achieved PR or SD after 4 doses could receive additional 2 doses of ASP7517 in combination with pembrolizumab. Subsequent to Treatment Period, all participants, except those with iCPD, iUPD who were not clinically stable or had clinical disease progression per independent central review/local review, entered the Observation Period were allowed to continue to receive pembrolizumab alone up to total of 17 doses of pembrolizumab to monitor treatment response and were followed for up to 96 weeks until iCPD, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the EOT visit, participants completed the Safety follow-up visits 30, 60 and 90 days.
- Phase 1:Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab: Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4 to 6 mL/minute) (1 Cycle=28 days) in combination with 400mg pembrolizumab infusion (over 30 minutes) with up to 4 doses every 6 weeks. Following first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (radiological response or SD/reduction of disease-related symptoms) continued further treatment with ASP7517 and pembrolizumab as decided by investigator. Participants who achieved confirmed CR within first 4 cycles could not receive further treatment with ASP7517 at cycle 5 and 6; and participants who achieved PR or SD after 4 doses could receive additional 2 doses of ASP7517 in combination with pembrolizumab. Subsequent to Treatment Period, all participants, except those with iCPD, iUPD who were not clinically stable or had clinical disease progression per independent central review or local review, entered Observation Period were allowed to continue to receive pembrolizumab alone up to total of 17 doses of pembrolizumab to monitor treatment response and were followed for up to 96 weeks until iCPD (confirmed by independent central review or local review), initiation of new anticancer therapy or meeting 1 of Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days.
Period: Phase 1 Dose Escalation (Up to 817 Days)
Arm/Group | Phase 1:Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2:Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1:Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1:Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Started | 3 | 8 | 0 | 3 | 8
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 3 | 8 | 0 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 4
Not completed — Progressive Disease | 3 | 4 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Period: Phase 2 Dose Expansion (Up to 504 Days)
Arm/Group | Phase 1:Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2:Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1:Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1:Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Started | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) consisted of all participants who took at least 1 dose of study drug.
Groups:
- Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose): Participants received one dose of ASP7517 1x10^7 cells/dose for up to 6 doses (168 days) by IV infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days). Following the first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (defined as radiological response or SD, or reduction of disease-related symptoms) continued further treatment with ASP7517, as decided by the investigator. After completing 4 cycles of treatment, any participants who achieved confirmed CR did not continue with ASP7517, and any participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD (per independent central review or local review) and who were not clinically stable or clinical progression was confirmed by the investigator and were followed for up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the EOT visit, participants completed the Safety follow-up visits 30, 60 and 90 days.
- Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose): Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) by IV infusion (4 to 6 mL/minute) on Day 1 of each cycle (1 Cycle=28 days).Following the first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (defined as radiological response or SD, or reduction of disease-related symptoms) continued further treatment with ASP7517, as decided by the investigator. After completing 4 cycles of treatment, any participants who achieved confirmed CR did not continue with ASP7517, and any participants who achieved PR or SD received an additional 2 doses. Participants entered an Observation Period except those with iCPD, iUPD (per independent central review or local review) and who were not clinically stable or clinical progression was confirmed by the investigator and were followed for up to 48 weeks until iCPD per independent central review, initiation of a new anticancer therapy or meeting 1 of the Observation Period discontinuation criteria, whichever occurred first. After the EOT visit, participants completed the Safety follow-up visits 30, 60 and 90 days.)
- Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab: Participants received ASP7517 1x10^7 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4 to 6 mL/minute) (1 Cycle=28 days) in combination with 400mg pembrolizumab infusion (over 30 minutes) with up to 4 doses every 6 weeks. Following first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (radiological response or SD/reduction of disease-related symptoms) continued further treatment with ASP7517 and pembrolizumab as decided by investigator. Participants who achieved confirmed CR within first 4 cycles could not receive further treatment with ASP7517 at cycle 5 and 6; and participants who achieved PR or SD after 4 doses could receive additional 2 doses of ASP7517 in combination with pembrolizumab. Subsequent to Treatment Period, all participants, except those with iCPD, iUPD who were not clinically stable or had clinical disease progression per independent central review or local review, entered Observation Period were allowed to continue to receive pembrolizumab alone up to total of 17 doses of pembrolizumab to monitor treatment response and were followed for up to 96 weeks until iCPD (confirmed by independent central review or local review), initiation of new anticancer therapy or meeting 1 of Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days.
- Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) and Pembrolizumab: Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4 to 6 mL/minute) (1 Cycle=28 days) in combination with 400mg pembrolizumab infusion (over 30 minutes) with up to 4 doses every 6 weeks. Following first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (radiological response or SD/reduction of disease-related symptoms) continued further treatment with ASP7517 and pembrolizumab as decided by investigator. Participants who achieved confirmed CR within first 4 cycles could not receive further treatment with ASP7517 at cycle 5 and 6; and participants who achieved PR or SD after 4 doses could receive additional 2 doses of ASP7517 in combination with pembrolizumab. Subsequent to Treatment Period, all participants, except those with iCPD, iUPD who were not clinically stable or had clinical disease progression per independent central review or local review, entered Observation Period were allowed to continue to receive pembrolizumab alone up to total of 17 doses of pembrolizumab to monitor treatment response and were followed for up to 96 weeks until iCPD (confirmed by independent central review or local review), initiation of new anticancer therapy or meeting 1 of Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) and Pembrolizumab | Total
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (16.3) | 51.6 (13.6) | 53.0 (12.7) | 61.3 (4.7) | 61.8 (12.1) | 58.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 1 | 2 | 3 | 13
  Male | 1 | 3 | 1 | 1 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 2 | 2 | 8 | 23
  Not Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 2
  White | 3 | 6 | 2 | 1 | 8 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: Participants] — ECOG Scale was used to assess performance status. Grades: 0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory, able to carry out work of light nature. 2: Ambulatory, capable of self-care, unable to carry out work activities. Up and about more than 50% waking hours. 3: Capable of limited self-care, confined to bed/chair more than 50% waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair. 5: Dead. Only participants with ECOG grades were reported.
  Participants
    Grade 0 | 1 | 4 | 2 | 1 | 3 | 11
    Grade 1 | 2 | 4 | 0 | 2 | 5 | 13
    Grade 2 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events: Monotherapy
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the study drug. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An AE was considered "serious" if, it resulted in any of the following outcomes: resulted in death; was life-threatening; resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; resulted in congenital anomaly, or birth defect; required inpatient hospitalization; or led to prolongation of hospitalization; other medically important events. A treatment-emergent adverse event (TEAE) was defined as an AE observed after the date of first dose until 30 days after the last dose.
Time Frame: From first dose up to 30 days after last dose (maximum treatment duration: approximately 534[504+30] days)
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose)
Number analyzed (Participants) | 3 | 8 | 2
Participants
  TEAEs | 3 | 7 | 2
  SAEs | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events: Combination Therapy
Description: as for outcome 1
Time Frame: From first dose up to 30 days after last dose (maximum treatment duration: approximately 847[817+30] days)
Population: SAF
Measure: Number; unit: Participants
Groups:
- Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab: Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4 to 6 mL/minute) (1 Cycle=28 days) in combination with 400mg pembrolizumab infusion (over 30 minutes) with up to 4 doses every 6 weeks. Following first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (radiological response or SD/reduction of disease-related symptoms) continued further treatment with ASP7517 and pembrolizumab as decided by investigator. Participants who achieved confirmed CR within first 4 cycles could not receive further treatment with ASP7517 at cycle 5 and 6; and participants who achieved PR or SD after 4 doses could receive additional 2 doses of ASP7517 in combination with pembrolizumab. Subsequent to Treatment Period, all participants, except those with iCPD, iUPD who were not clinically stable or had clinical disease progression per independent central review or local review, entered Observation Period were allowed to continue to receive pembrolizumab alone up to total of 17 doses of pembrolizumab to monitor treatment response and were followed for up to 96 weeks until iCPD (confirmed by independent central review or local review), initiation of new anticancer therapy or meeting 1 of Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days.
Arm/Group | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8
Participants
  TEAEs | 3 | 8
  SAEs | 1 | 2

3. Primary Outcome: Number of Participants With ECOG Performance Status at Cycle (C) 1 Day (D) 1
Description: The ECOG Scale was used to assess performance status. Grade Description: 0 - Fully active, able to carry on all pre disease performance without restriction. 1 - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. 2 - Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. 5 -Dead.
Time Frame: At C1D1
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
Participants
  Grade 0 | 1 | 4 | 2 | 1 | 3
  Grade 1 | 2 | 4 | 0 | 2 | 5
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With ECOG Performance Status at C1D2
Description: as for outcome 3
Time Frame: At C1D2
Population: SAF with available data was analyzed. As per protocol no participants were planned to be enrolled in C1D2 for monotherapy dose expansion therefore, no participants were included in this arm.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 0 | 3 | 8
Participants
  Grade 0 | 1 | 3 |  | 1 | 3
  Grade 1 | 2 | 5 |  | 2 | 3
  Grade 2 | 0 | 0 |  | 0 | 2
  Grade 3 | 0 | 0 |  | 0 | 0
  Grade 4 | 0 | 0 |  | 0 | 0
  Grade 5 | 0 | 0 |  | 0 | 0

5. Primary Outcome: Number of Participants With ECOG Performance Status at C1D4
Description: as for outcome 3
Time Frame: At C1D4
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
Participants
  Grade 0 | 1 | 4 | 1 | 1 | 3
  Grade 1 | 2 | 4 | 1 | 2 | 3
  Grade 2 | 0 | 0 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With ECOG Performance Status at C1D8
Description: as for outcome 3
Time Frame: At C1D8
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
Participants
  Grade 0 | 1 | 3 | 1 | 1 | 3
  Grade 1 | 2 | 5 | 1 | 2 | 4
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With ECOG Performance Status at C1D15
Description: as for outcome 3
Time Frame: At C1D15
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
Participants
  Grade 0 | 1 | 3 | 1 | 1 | 2
  Grade 1 | 2 | 5 | 1 | 2 | 5
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With ECOG Performance Status at C2D1
Description: as for outcome 3
Time Frame: At C2D1
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 2 | 7 | 2 | 3 | 7
Participants
  Grade 0 | 0 | 3 | 1 | 2 | 2
  Grade 1 | 2 | 4 | 1 | 1 | 4
  Grade 2 | 0 | 0 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With ECOG Performance Status at C2D4
Description: as for outcome 3
Time Frame: At C2D4
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 2 | 6 | 2 | 3 | 6
Participants
  Grade 0 | 0 | 3 | 1 | 2 | 1
  Grade 1 | 2 | 3 | 1 | 1 | 5
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With ECOG Performance Status at C2D8
Description: as for outcome 3
Time Frame: At C2D8
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 2 | 5 | 2 | 3 | 7
Participants
  Grade 0 | 0 | 2 | 1 | 2 | 1
  Grade 1 | 2 | 3 | 1 | 1 | 5
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With ECOG Performance Status at C2D15
Description: as for outcome 3
Time Frame: At C2D15
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 2 | 5 | 2 | 3 | 6
Participants
  Grade 0 | 0 | 1 | 0 | 2 | 1
  Grade 1 | 2 | 4 | 2 | 1 | 5
  Grade 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With ECOG Performance Status at C3D1
Description: as for outcome 3
Time Frame: At C3D1
Population: SAF with available data was analyzed. No participants from Phase 2 monotherapy dose expansion entered C3D1 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 3 | 0 | 1 | 5
Participants
  Grade 0 | 0 | 1 |  | 1 | 1
  Grade 1 | 1 | 2 |  | 0 | 4
  Grade 2 | 0 | 0 |  | 0 | 0
  Grade 3 | 0 | 0 |  | 0 | 0
  Grade 4 | 0 | 0 |  | 0 | 0
  Grade 5 | 0 | 0 |  | 0 | 0

13. Primary Outcome: Number of Participants With ECOG Performance Status at C3D8
Description: as for outcome 3
Time Frame: At C3D8
Population: SAF with available data was analyzed. No participants from Phase 2 monotherapy dose expansion entered C3D8 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 3 | 0 | 1 | 5
Participants
  Grade 0 | 0 | 1 |  | 1 | 1
  Grade 1 | 1 | 2 |  | 0 | 4
  Grade 2 | 0 | 0 |  | 0 | 0
  Grade 3 | 0 | 0 |  | 0 | 0
  Grade 4 | 0 | 0 |  | 0 | 0
  Grade 5 | 0 | 0 |  | 0 | 0

14. Primary Outcome: Number of Participants With ECOG Performance Status at C3D15
Description: as for outcome 3
Time Frame: At C3D15
Population: SAF with available data was analyzed. No participants from Phase 2 monotherapy dose expansion entered C3D15 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 2 | 0 | 1 | 5
Participants
  Grade 0 | 0 | 0 |  | 1 | 1
  Grade 1 | 1 | 2 |  | 0 | 4
  Grade 2 | 0 | 0 |  | 0 | 0
  Grade 3 | 0 | 0 |  | 0 | 0
  Grade 4 | 0 | 0 |  | 0 | 0
  Grade 5 | 0 | 0 |  | 0 | 0

15. Primary Outcome: Number of Participants With ECOG Performance Status at C4D1
Description: as for outcome 3
Time Frame: At C4D1
Population: SAF with available data was analyzed. No participants from Phase 2 monotherapy dose expansion entered C4D1 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 2 | 0 | 1 | 4
Participants
  Grade 0 | 0 | 0 |  | 1 | 1
  Grade 1 | 1 | 2 |  | 0 | 3
  Grade 2 | 0 | 0 |  | 0 | 0
  Grade 3 | 0 | 0 |  | 0 | 0
  Grade 4 | 0 | 0 |  | 0 | 0
  Grade 5 | 0 | 0 |  | 0 | 0

16. Primary Outcome: Number of Participants With ECOG Performance Status at C4D8
Description: as for outcome 3
Time Frame: At C4D8
Population: SAF with available data was analyzed. No participants from Phase 2 monotherapy dose expansion entered C4D8 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 4
Participants
  Grade 0 | 0 | 0 |  | 1 | 1
  Grade 1 | 1 | 0 |  | 0 | 3
  Grade 2 | 0 | 0 |  | 0 | 0
  Grade 3 | 0 | 1 |  | 0 | 0
  Grade 4 | 0 | 0 |  | 0 | 0
  Grade 5 | 0 | 0 |  | 0 | 0

17. Primary Outcome: Number of Participants With ECOG Performance Status at C4D15
Description: as for outcome 3
Time Frame: At C4D15
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation (with dosage ASP7517 1x10^8 cells/dose) and Phase 2 monotherapy dose expansion entered C4D15 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 3
Participants
  Grade 0 | 0 |  |  | 1 | 0
  Grade 1 | 1 |  |  | 0 | 3
  Grade 2 | 0 |  |  | 0 | 0
  Grade 3 | 0 |  |  | 0 | 0
  Grade 4 | 0 |  |  | 0 | 0
  Grade 5 | 0 |  |  | 0 | 0

18. Primary Outcome: Number of Participants With ECOG Performance Status at C5D1
Description: as for outcome 3
Time Frame: At C5D1
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation, Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered C5D1 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 3
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

19. Primary Outcome: Number of Participants With ECOG Performance Status at C5D8
Description: as for outcome 3
Time Frame: At C5D8
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation, Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered C5D8 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 3
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

20. Primary Outcome: Number of Participants With ECOG Performance Status at C5D15
Description: as for outcome 3
Time Frame: At C5D15
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation, Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered C5D15 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 3
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

21. Primary Outcome: Number of Participants With ECOG Performance Status at C6D1
Description: as for outcome 3
Time Frame: At C6D1
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation, Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered C6D1 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
Participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 3
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

22. Primary Outcome: Number of Participants With ECOG Performance Status at C6D8
Description: as for outcome 3
Time Frame: At C6D8
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation, Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered C6D8 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
Participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 2
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

23. Primary Outcome: Number of Participants With ECOG Performance Status at C6D15
Description: as for outcome 3
Time Frame: At C6D15
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation, Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered C6D15 therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
Participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 1
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

24. Primary Outcome: Number of Participants With ECOG Performance Status at End of Treatment (EOT): Monotherapy
Description: The ECOG Scale was used to assess performance status. Grade Description: 0 - Fully active, able to carry on all pre disease performance without restriction. 1 - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. 2 - Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. 5 -Dead. EOT visit was conducted for all participants after 7 days of last dose.
Time Frame: At EOT (Approximately 511 [504 +7] days)
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose)
Number analyzed (Participants) | 2 | 7 | 2
Participants
  Grade 0 | 1 | 2 | 0
  Grade 1 | 1 | 1 | 2
  Grade 2 | 0 | 2 | 0
  Grade 3 | 0 | 2 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

25. Primary Outcome: Number of Participants With ECOG Performance Status at End of Treatment (EOT): Combination Therapy.
Description: as for outcome 24
Time Frame: At EOT (Approximately 824 [817 +7] days)
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 5
Participants
  Grade 0 | 0 | 1
  Grade 1 | 1 | 4
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

26. Primary Outcome: Number of Participants With ECOG Performance Status at 30 Day Follow Up: Monotherapy
Description: as for outcome 3
Time Frame: At 30 days safety Follow Up (Approximately 541 [511+30] days)
Population: SAF with available data was analyzed. No participants from Phase 1 monotherapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered the 30 day follow up period therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose)
Number analyzed (Participants) | 0 | 1 | 0
Participants
  Grade 0 |  | 0 |
  Grade 1 |  | 0 |
  Grade 2 |  | 1 |
  Grade 3 |  | 0 |
  Grade 4 |  | 0 |
  Grade 5 |  | 0 |

27. Primary Outcome: Number of Participants With ECOG Performance Status at 30 Day Follow Up: Combination Therapy
Description: as for outcome 3
Time Frame: At 30 days safety Follow Up (Approximately 854 [824+30 ] days)
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 1 | 3
Participants
  Grade 0 | 1 | 1
  Grade 1 | 0 | 2
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

28. Primary Outcome: Number of Participants With ECOG Performance Status at 60 Day Follow Up: Monotherapy
Description: as for outcome 3
Time Frame: At 60 days safety Follow Up (Approximately 571 [511+60] days)
Population: SAF with available data was analyzed.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose)
Number analyzed (Participants) | 1 | 1 | 1
Participants
  Grade 0 | 0 | 1 | 0
  Grade 1 | 1 | 0 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

29. Primary Outcome: Number of Participants With ECOG Performance Status at 60 Day Follow Up: Combination Therapy
Description: as for outcome 3
Time Frame: At 60 days safety Follow Up (Approximately 884 [824+60] days)
Population: SAF with available data was analyzed. No participants from Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) entered the 60 day follow up period therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 1
Participants
  Grade 0 |  | 0
  Grade 1 |  | 1
  Grade 2 |  | 0
  Grade 3 |  | 0
  Grade 4 |  | 0
  Grade 5 |  | 0

30. Primary Outcome: Number of Participants With ECOG Performance Status at 90 Day Follow Up: Monotherapy
Description: as for outcome 3
Time Frame: At 90 days safety follow up (Approximately 601 [511+90] days)
Population: SAF with available data was analyzed. No participants from the Phase 1 monotherapy therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) and Phase 2 monotherapy dose expansion entered the 90 day follow up period therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose)
Number analyzed (Participants) | 0 | 1 | 0
Participants
  Grade 0 |  | 1 |
  Grade 1 |  | 0 |
  Grade 2 |  | 0 |
  Grade 3 |  | 0 |
  Grade 4 |  | 0 |
  Grade 5 |  | 0 |

31. Primary Outcome: Number of Participants With ECOG Performance Status at 90 Day Follow Up: Combination Therapy
Description: as for outcome 3
Time Frame: At 90 days safety follow up (Approximately 914 [824+90] days)
Population: SAF with available data was analyzed. No participants from the Phase 1 combination therapy dose escalation (with dosage ASP7517 1x10^7 cells/dose) entered the 90 day follow up period therefore, the number of participants is 0.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 1
Participants
  Grade 0 |  | 0
  Grade 1 |  | 1
  Grade 2 |  | 0
  Grade 3 |  | 0
  Grade 4 |  | 0
  Grade 5 |  | 0

32. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT: any event occurring within 28 days of first dose on C1D1 and graded as: *Non-hematologic AEs >= grade 3 and not resolving to <= grade 2 within 72 hours. *Confirmed Hy's law case. *Infusion-related reactions requiring infusion discontinuation, prolonged delay (> 2 weeks) in initiating C2 due to treatment-related toxicity. *Any treatment-related toxicity causing discontinuation in C1. *Grade >= 3 thrombocytopenia/bleeding requiring transfusion/hospitalization, grade >= 3 anemia requiring transfusion, grade 3 febrile neutropenia with/without infection and grade 5 treatment-related toxicity, grade >= 2 pneumonitis, grade >= 2 encephalopathy, meningitis or motor/sensory neuropathy. *Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) > 5 × upper limit of normal (ULN) in participants without liver metastases, AST/ALT > 8×ULN in participants with liver metastases, total bilirubin > 3×ULN (grade >= 3). *Guillain-Barré syndrome/myasthenic syndrome/myasthenia gravis.
Time Frame: From C1D1 up to C1D28
Population: The DLT evaluation analysis set (DEAS) consisted of all participants in SAF excluding participants who met any of the following criteria:
  * Participant was discovered to have enrolled without fully satisfying eligibility criteria.
  * Participant received less than the planned dose in cycle 1 for reasons other than DLT.
  * Participant had no DLT and withdraws from the study before the end of DLT evaluation period.
  DLTs were analyzed only in Phase 1 .
Measure: Number; unit: Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 8
Participants | 0 | 0 | 0 | 0

33. Primary Outcome: Objective Response Rate (iORR) Per Immune Response Evaluation Criteria in Solid Tumors (iRECIST) by Investigator Assessment
Description: iORR was defined as the percentage of participants for each dose level whose best overall response was rated as confirmed iCR or iPR per iRECIST by independent central review. iCR was complete response based on iRECIST and defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR was partial response based on iRECIST was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
  iORR assessments included:
  * iORR with confirmed response by investigator assessment
  * iORR with unconfirmed response by investigator assessment For confirmed response for iCR/iPR, scan had to be done 4 weeks after iPR/iCR was first observed. Participants who had iCR/iPR were considered as having confirmed response and those that did not fulfil this criteria were considered as having unconfirmed response.
Time Frame: From first dose up to 954 days
Population: Response analysis set (RAS) consisted of all participants who were enrolled and received at least 1 dose of investigational product (IP) and had at least 1 postbaseline primary efficacy measurement.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 7
Percentage of Participants
  iORR with confirmation | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0]
  iORR without confirmation | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0]

34. Secondary Outcome: Objective Response Rate (ORR) Per RECIST v1.1 by Investigator Assessment
Description: ORR was defined as the percentage of participants for each dose level whose best overall response is rated as complete response (CR) or partial response (PR) per RECIST v1.1. CR was complete response based on RECIST and defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 mm in the short axis. PR was partial response based on RECIST and defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
  ORR assessment included:
  * ORR with confirmed response by investigator assessment
  * ORR with unconfirmed response by investigator assessment For confirmed response for CR/PR, scan had to be done 4 weeks after PR/CR was first observed. Participants who had CR/PR were considered as having confirmed response and those that did not fulfil this criteria were considered as having unconfirmed response.
Time Frame: From first dose up to 954 days
Population: RAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 7
Percentage of Participants
  ORR with confirmation | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0]
  ORR without confirmation | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0]

35. Secondary Outcome: Disease Control Rate Per iRECIST (iDCR) by Investigator Assessment
Description: iDCR: Percentage of participants for each dose level whose best overall response is rated as confirmed iCR, iPR or iSD per iRECIST. iCR: Complete response based on iRECIST, defined as disappearance of all target/non target lesions and pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR: Partial response based on iRECIST, defined as at least 30% decrease in the sum of diameters of target lesions, with reference to the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for iPR nor sufficient increase to qualify for PD. PD: Defined as at least 20% increase in the sum of diameters of target lesions, with reference to the smallest sum of diameters recorded since the treatment started. For confirmed response for iCR/iPR, scan had to be done 4 weeks after iPR/iCR was first observed. Participants who had iCR/iPR were considered as having confirmed response and those that did not fulfil this criteria were considered as having unconfirmed response.
Time Frame: From first dose up to 954 days
Population: RAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 7
Percentage of Participants
  iDCR with confirmation | 33.3 [0.8 to 90.6] | 42.9 [9.9 to 81.6] | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 57.1 [18.4 to 90.1]
  iDCR without confirmation | 33.3 [0.8 to 90.6] | 42.9 [9.9 to 81.6] | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 57.1 [18.4 to 90.1]

36. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 by Investigator Assessment
Description: DCR: Percentage of participants for each dose level whose best overall response is rated as confirmed CR, PR or SD per RECIST v1.1. CR: Complete response based on RECIST and defined as disappearance of all target/non target lesions and any pathological lymph nodes must be <10 mm in the short axis. PR: Partial response based on RECIST and defined as at least a 30% decrease in the sum of diameters of target lesions, with reference to, the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for iPR nor sufficient increase to qualify for PD. PD: At least a 20% increase in the sum of diameters of target lesions, with reference to, the smallest sum of diameters recorded since treatment started. For confirmed response for CR/PR, scan had to be done 4 weeks after PR/CR was first observed. Participants who had CR/PR were considered as having confirmed response and those that did not fulfil this criteria were considered as having unconfirmed response.
Time Frame: From first dose up to 954 days
Population: RAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose); Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab: Participants received ASP7517 1x10^8 cells/dose for up to 6 doses (168 days) on Day 1 of each cycle by IV infusion (4 to 6 mL/minute) (1 Cycle=28 days) in combination with 400mg pembrolizumab infusion (over 30 minutes) with up to 4 doses every 6 weeks. Following first 2 cycles, participants who had not met any individual treatment discontinuation criteria and were receiving clinical benefit (radiological response or SD/reduction of disease-related symptoms) continued further treatment with ASP7517 and pembrolizumab as decided by investigator. Participants who achieved confirmed CR within first 4 cycles could not receive further treatment with ASP7517 at cycle 5 and 6; and participants who achieved PR or SD after 4 doses could receive additional 2 doses of ASP7517 in combination with pembrolizumab. Subsequent to Treatment Period, all participants, except those with iCPD, iUPD who were not clinically stable or had clinical disease progression per independent central review or local review, entered Observation Period were allowed to continue to receive pembrolizumab alone up to total of 17 doses of pembrolizumab to monitor treatment response and were followed for up to 96 weeks until iCPD (confirmed by independent central review or local review), initiation of new anticancer therapy or meeting 1 of Observation Period discontinuation criteria, whichever occurred first. After EOT visit, participants completed Safety follow-up visits 30, 60 and 90 days.
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 7
Percentage of Participants
  DCR with confirmation | 33.3 [0.8 to 90.6] | 42.9 [9.9 to 81.6] | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 57.1 [18.4 to 90.1]
  DCR without confirmation | 33.3 [0.8 to 90.6] | 42.9 [9.9 to 81.6] | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 57.1 [18.4 to 90.1]

37. Secondary Outcome: Progression-Free Survival Per iRECIST (iPFS) Using Investigator Assessment
Description: iPFS was defined as the time from the start of the study treatment until death from any cause or radiographic disease progression assessed per iRECIST by independent central review and investigator assessment, whichever occurs first. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started. Kaplan Meier estimate was used for analysis of time-to-event endpoints.
Time Frame: From first dose until death from any cause or radiographic disease progression (up to 954 days)
Population: Full analysis set (FAS) consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
days | 398.0 [57.0 to 404.0] | 57.0 [32.0 to 112.0] | 77.0 [NA to NA] — Due to low number of events, lower and upper limit of CI was not estimable. | 106.0 [54.0 to 142.0] | 106.0 [37.0 to 164.0]

38. Secondary Outcome: Progression-Free Survival Per RECIST (PFS) Using Investigator Assessment
Description: PFS was defined as the time from the start of the study treatment until death from any cause or radiographic disease progression assessed per RECIST by independent central review and investigator assessment, whichever occurred first. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started. Kaplan Meier estimate was used for analysis of time-to-event endpoints.
Time Frame: From first dose until death from any cause or radiographic disease progression (up to 954 days)
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
days | 57.0 [29.0 to 99.0] | 57.0 [32.0 to 112.0] | 77.0 [NA to NA] — Due to low number of events, lower and upper limit of CI was not estimable. | 57.0 [29.0 to 99.0] | 57.0 [32.0 to 112.0]

39. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose until the date of death from any cause (death date - first dose date + 1). For a participant who is not known to have died by the end of study follow-up, OS is censored at the date of last contact (date of last contact - first dose date + 1). Kaplan Meier estimate was used for analysis of time-to-event endpoints.
Time Frame: From first dose until death from any cause (up to 954 days)
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 3 | 8 | 2 | 3 | 8
days | 404.0 [398.0 to NA] — Due to low number of events, upper limit of CI was not estimable. | 169.0 [57.0 to 297.0] | NA [77.0 to NA] — Due to low number of events, median and upper limit of CI was not estimable. | NA [142.0 to NA] — Due to low number of events, median and upper limit of CI was not estimable. | NA [200.0 to NA] — Due to low number of events, median and upper limit of CI was not estimable.

40. Secondary Outcome: Duration of Response Per iRECIST (iDOR)
Description: iDOR was defined as the time from the date of the first response iCR/iPR (whichever was first recorded) to the date of radiographical progression or date of censoring. iCR was complete response based on iRECIST and defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR was partial response based on iRECIST was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: From first response up to the date of radiographical progression (up to 954 days)
Population: No participant had a response of iCR or iPR and therefore iDOR was not evaluable.
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1
Description: DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression or date of censoring. DOR will be calculated only for the subgroup of participants with confirmed response CR/PR per RECIST v1.1, separately for independent central review and for investigator assessment. CR was complete response based on RECIST and defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 mm in the short axis. PR was partial response based on RECIST and defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: From first response up to the date of radiographical progression (up to 954 days)
Population: No participant had a response of CR or PR and therefore DOR was not evaluable.
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8cells/Dose) and Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time frame for adverse events: From first dose up to 30 days after last dose (approximately 534 days for monotherapy and approximately 847 days for combination therapy). Time frame for all-cause mortality: From randomization up to end of study (approximately 954 days)
Description: All-cause mortality: All randomized participants. Adverse events: SAF consisted of all participants who took at least 1 dose of study drug.
Arm/Group | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/8 | 1/2 | 1/3 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/8 | 0/2 | 1/3 | 2/8
Other Adverse Events (participants affected / at risk) | 3/3 | 7/8 | 2/2 | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) (N=3) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) (N=8) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) (N=2) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab (N=3) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) and Pembrolizumab (N=8)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) (N=3) | Phase 1: Monotherapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) (N=8) | Phase 2: Monotherapy Dose Expansion (ASP7517 1x10^8 Cells/Dose) (N=2) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^7 Cells/Dose) and Pembrolizumab (N=3) | Phase 1: Combination Therapy Dose Escalation (ASP7517 1x10^8 Cells/Dose) and Pembrolizumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (3) | 1 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Catheter site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (6) | 2 (2) | 2 (2) | 4 (5)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04837196/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT04837196/SAP_001.pdf